CLINICAL TRIAL: NCT05103280
Title: Improving Walking in Peripheral Artery Disease Using Specially Designed Assistive Shoes
Brief Title: Improving Walking in Peripheral Artery Disease
Acronym: PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F3877-P; I21RX003877 (NIH)
Record Dates: First submitted 2021-10-19; First posted 2021-11-02 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral artery disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: Ten patients will wear assistive shoes for 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Progressive improvement in walking performance (Experimental): A total of ten patients with peripheral artery disease will be enrolled for this arm and wear the assistive tennis shoes for three-months as an intervention.
  Interventions: Other: Assistive tennis shoes

INTERVENTIONS:
Other: Assistive tennis shoes — Assistive shoes include carbon-fiber and spring loaded shoes.

SUMMARY:
Peripheral artery disease (PAD) is a cardiovascular disease manifesting from systemic atherosclerosis that blocks the leg arteries and results in insufficient blood flow to the lower extremities. Limb ischemia from PAD is the most common disorder treated within the vascular surgical service of the Omaha Veterans Affairs Medical Center. PAD also accounts for one-third of the operations performed in the VA Medical Centers nationwide. The risk of mortality of Veterans with PAD is substantial; nearly 30% of Veterans with PAD died within 3.8 years of diagnosis. This project aims to establish the feasibility and acceptability of specially designed assistive shoes in patients with PAD and to determine if there are any potential benefits of using these shoes over standard shoes. These assistive shoes may enable patients to carry out desired activities of daily living with less pain and more physical activity. Increasing physical activity will decrease morbidity and mortality. If proven beneficial, the findings will lead to a novel and conservative rehabilitation protocol that directly benefits Veterans nationwide.

DETAILED DESCRIPTION:
The long-term goal of this project is to improve mobility, functional independence, and quality of life in patients with peripheral artery disease (PAD) by using specially designed assistive shoes. PAD is a manifestation of systemic atherosclerosis, producing blockages in the leg arteries, resulting in insufficient blood flow to the lower extremities. Limb ischemia from PAD is the most common disorder treated within the vascular surgical service of the Omaha Veterans Affairs Medical Center. PAD also accounts for one-third of the operations performed nationwide in the VA. Walking-induced muscle pain, known as intermittent claudication, is the most common PAD symptom. Claudicating patients with PAD walk slower, have reduced quality of life and lose independence in performing activities of daily living. The investigators have identified consistent deficits of the ankle plantarflexors to effectively push-off during walking. Currently, there is a critical treatment gap for patients whose disease presentation does not warrant an operative approach, but who desire to restore their functional independence and walking ability. Specially designed assistive shoes (carbon fiber: CF; spring-loaded: SL) with specific mechanical properties to absorb and release energy, have been shown to promote push-off efficiency in walkers and runners. These shoes may lead to improved push-off in populations with reduced ankle push-off capacity, but this has not been tested yet. This work proposes to evaluate patient preferences in terms of using assistive shoes and whether these shoes improve walking performance in claudicating patients with PAD. The investigators hypothesize that using assistive shoes (either CF or SL, based on their preference) for three months will lead to improved walking performance in patients with PAD. The investigators also hypothesize that the subject-reported preference of assistive shoes (CF versus SL) will be positive based on comfort, fatigue, ease of walking, and feasibility at the baseline session. Two hypotheses will be tested by the following three specific aims:

Aim 1: Determine the subject-reported preference of assistive shoes at the Baseline visit.

Aim 2: Determine the progressive improvements in physical activity, quality of life, and walking distance after a three-month assistive shoe intervention.

Twenty patients with PAD will be recruited. Aim 1 will primarily focus on qualitative measurements of subjects' reported preferences to identify which assistive shoes are feasible for patients with PAD to use during the three months of intervention. Visual-analog scales, rate of perceived exertion, and interviews will be used to assess comfort, fatigue, intensity, and feasibility after each shoe condition of Aim 1. Patients will wear the preferred assistive shoes of their choice for regular daily use for three months as a conservative intervention. Physical activity, quality of life, and walking distances will be assessed prior to the start of the intervention and after three months of intervention. Overall, the aims will demonstrate the feasibility and acceptability of assistive shoes in patients with PAD. Results will support a full clinical trial and guide necessary intervention length and potential rehabilitation recommendations.

ELIGIBILITY:
Inclusion Criteria:

At entry into the study, all patients must:

* be able to give written, informed consent
* demonstrate positive history of chronic claudication
* have an ankle brachial index < 0.90 at rest
* have a stable blood pressure regimen, stable lipid regimen, stable diabetes regimen and risk factor control for 6 weeks

Exclusion Criteria:

Any potential subjects will be excluded if they have:

* rest pain or tissue loss due to peripheral artery disease (Fontaine stage III and IV)
* acute lower extremity ischemic event secondary to thromboembolic disease or acute trauma
* walking capacity significantly limited by conditions other than claudication including leg (joint/musculoskeletal, neurologic) and systemic (heart, lung disease) pathology

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara A. Myers, PhD, Principal Investigator — Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE
Locations (1):
- Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created for sharing purposes. All the outcomes and results will be published in peer-reviewed journals and conference proceedings. The raw data will be shared in a de identified, anonymized dataset upon request with a written agreement from recipient. Therefore, the recipient will be able to complete follow-up and perform new analyses of the raw data.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The de-identified, anonymized dataset will only be shared after the completion of the study and publishing the outcomes in peer-reviewed journals and conference proceedings.

RESULTS

PARTICIPANT FLOW:
Groups:
- Progressive Improvement in Walking Performance: A total of 10 participants with peripheral artery disease were enrolled in this single-arm study. Each participant wore only one type of preferred assistive shoes-carbon-fiber insole shoes, or spring-loaded shoes-over the course of a three-month intervention period. The aim was to assess how walking performance changed within each participant following the use of assistive shoes, relative to their baseline performance.
Period: Overall Study
Arm/Group | Progressive Improvement in Walking Performance
Started | 10
SL for Intervention | 7
CF for Intervention | 3
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Progressive Improvement in Walking Performance
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (8.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Progressive improvement in walking performance: Female | 0
  Progressive improvement in walking performance: Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Changes in Walking Distance After Three-months Intervention
Description: In this single-arm study, investigators assessed absolute claudication walking distance using the Gardner treadmill test while participants walked in their normal footwear. This assessment was conducted both before and after a three-month intervention using assistive shoes-either carbon fiber or spring-loaded-selected based on participant preference. No control group was included.
Time Frame: Baseline and after three-months intervention
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Progressive Improvement in Walking Performance
Number analyzed (Participants) | 10
meters
  Baseline | 289.68 (196.11)
  After Three months | 262.95 (165.97)

2. Primary Outcome: Comfort Level of Wearing Assistive Shoe Expressed as a Numeric Value and This Value Will be Rated by Participants
Description: At the baseline session, participants will be asked to rate the comfort of each assistive shoe on a scale from 0 to 10, where 0 indicates "Low comfort" and 10 indicates "High comfort." During this session, all participants will walk in three different shoes and provide a comfort rating for each. Based on these ratings, one shoe will be selected for the participant to use over the following three months.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Progressive Improvement in Walking Performance
Number analyzed (Participants) | 10
units on a scale
  standard shoe | 5.5 (1.08)
  carbon fiber | 5.9 (2.3)
  spring loaded | 6.6 (2.06)

3. Secondary Outcome: Changes in Vertical Ground Reaction Force After Three-months Intervention
Description: In this single-arm study, investigators assessed vertical ground reaction force from a pressure-instrumented treadmill during the Gardner treadmill test while walking in their normal shoes. This assessment was conducted both before and after a three-month intervention using assistive shoes-either carbon fiber or spring-loaded-selected based on participant preference. No control group was included.
Time Frame: Baseline and after three-months intervention
Measure: Mean (Standard Deviation); unit: Newton
Groups:
- Ground Reaction Force Improvement: Ground reaction forces will be measured at Baseline and after three months of using assistive shoes.
Arm/Group | Ground Reaction Force Improvement
Number analyzed (Participants) | 10
Newton
  Baseline | 769.34 (150.09)
  after three-months intervention | 845.38 (118.24)

4. Secondary Outcome: Changes in Muscle Oxygenation After Three-months Intervention
Description: In this single-arm study, investigators will assess minimum muscle oxygenation during the Gardner treadmill test while wearing their normal shoes.
  This assessment was conducted both before and after a three-month intervention using assistive shoes-either carbon fiber or spring-loaded-selected based on participant preference. No control group was included.
Time Frame: Baseline and after three-months intervention
Measure: Mean (Standard Deviation); unit: Muscle oxygen saturation percentage
Arm/Group | Ground Reaction Force Improvement
Number analyzed (Participants) | 10
Muscle oxygen saturation percentage
  Baseline | 36.82 (15.92)
  After three months | 40.02 (12.30)

5. Secondary Outcome: Changes in Physical Activity After Three-months Intervention
Description: In this single-arm study, investigators calculated the average number of steps per day as a measure of physical activity using an ActiGraph accelerometer worn by participants. All participants underwent a three-month intervention using assistive shoes-either carbon fiber or spring-loaded-selected based on their personal preference. No control group was included. Participants wore the accelerometer for 7 days before the intervention and again for 7 days after completing the three-month intervention period.
Time Frame: Baseline and after three-months intervention
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | Ground Reaction Force Improvement
Number analyzed (Participants) | 10
steps/day
  Baseline | 4099.102 (4035.33)
  After three months intervention | 4740.85 (4913.19)

6. Secondary Outcome: Changes in Rate of Perceived Exertion Score After Three-months Intervention
Description: In this single-arm study, investigators assessed the rate of perceived exertion (RPE) immediately after the Gardner treadmill test while participants walked in their normal footwear. This assessment was conducted both before and after a three-month intervention using assistive shoes-either carbon fiber or spring-loaded-selected based on participant preference. No control group was included. The RPE score ranged from 6 to 20, where 6 indicated no exertion at all and 20 indicated maximal exertion.
Time Frame: Baseline and after three-months intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Rate of Perceived Exertion in Progressive Treadmill Test Before and After Intervention: Patients will rate of perceived exertion score after a progressive treadmill test when walking with their normal shoes. The score ranges from six to twenty. Zero represents no exertion at all, and twenty represents maximal exertion.
Arm/Group | Rate of Perceived Exertion in Progressive Treadmill Test Before and After Intervention
Number analyzed (Participants) | 10
score on a scale
  Baseline | 12.6 (2.7)
  After three months | 13.25 (2.3)

ADVERSE EVENTS:
Time Frame: Baseline and three months after intervention.
Description: Adverse events were monitored throughout the study. Data collection followed the ClinicalTrials.gov definitions for adverse and serious adverse events. No alternative definitions were used. Participants were assessed for adverse events at baseline and again three months after the intervention.
Groups:
- Assistive Shoe Intervention for PAD Patients: Participants with peripheral artery disease (PAD) received an assistive shoe intervention designed to improve walking ability and reduce claudication symptoms. The shoes were tailored to support gait mechanics and enhance comfort during walking. Functional outcomes were assessed at baseline and again three months after the intervention.
Arm/Group | Assistive Shoe Intervention for PAD Patients
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT05103280/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/80/NCT05103280/ICF_000.pdf